CLINICAL TRIAL: NCT05652348
Title: Response Prediction of Hyperthermic Intraperitoneal Chemotherapy in Gastro- Intestinal Cancer
Acronym: Hi-STEP1
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: VTG-12
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Gastric Cancer; Colon Cancer; Peritoneal Carcinomatosis
Keywords: Organoid
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms; Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of tumor taken during standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Establishment of organoid cultures and in vitro sensitivity testing — Generating patient-derived tumor organoid models as well as orthotopic mouse models from peritoneal carcinomatosis lesions and to investigate their response to different therapies.

SUMMARY:
Patients with gastric or colon cancer with peritoneal carcinomatosis will receive a biopsy of the tumor during their primary curative surgery. The operation is performed according to standard and includes resection of the primary tumor and any metastases and followed by HIPEC (Intraperitoneal hyperthermic chemoperfusion) according to the respective hospital standard. Organoid cultures from the biopsies are established in the research laboratory.

Various chemotherapeutic agents are tested on these tumor organoids in the laboratory and the tumor organoids are analyzed in detail with regard to genetic alterations in order to find alterations that can be addressed, if necessary, by means of targeted drugs against peritoneal carcinomatosis.

ELIGIBILITY:
Inclusion Criteria:

* (Suspected) synchronous or metachronous peritoneal metastasis of adenocarcinoma of the stomach / gastroesophageal junction (GEJ) or of the colon or rectum
* intraoperative histological confirmation of synchronous or metachronous peritoneal carcinomatosis in gastric carcinoma (incl. GEJ) or colon carcinoma (incl. rectal carcinoma)
* Intraoperative peritoneal cancer index (PCI) ≤ 15 for gastric carcinoma and ≤ 20 for colon carcinoma.
* Possibility of surgical resection of peritoneal carcinomatosis (cytoreductive surgery) in curative intention with achievement of a Completeness of Cytoreduction Score (CCS) of 0-1
* No contraindication to surgery
* No contraindication against the performance of HIPEC
* Expected survival of 6 months at least
* ECOG ≤ 2
* Female and male patients ≥ 18 years of age
* Patient is able and willing to give written informed consent and comply with the study protocol

Exclusion Criteria:

* Presence of non-resectable distant metastases
* Patients with extensive metastasis (e.g., multiple bilobular liver metastases, hepatic and pulmonary metastases, multiple retroperitoneal lymph node metastases; oligometastasis is allowed)
* Patients with recurrence of peritoneal carcinomatosis (e.g., previous peritonectomy in the course of primary tumor resection)
* Patients after previous palliative chemotherapy or radiation of the tumor (exception: neoadjuvant and/or adjuvant therapies)
* Hypersensitivity/allergy to components of the planned intraperitoneal chemotherapy
* Patients not eligible for surgery/HIPEC (e.g., heart failure NYHA ≥III, myocardial infarction within the last 3 months before surgery, high-risk cardiac arrhythmias)
* Secondary malignant disease that occurred <5 years ago (exception: early stage of a localized tumor with in-sano resection, for example in situ carcinoma of the cervix, Adequately treated basal cell carcinoma of the skin)
* Patients who are housed in a closed facility
* Pregnant or breastfeeding patients, or patients who plan to become pregnant within 7 Months after the end of treatment to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are recruited consecutively during of the initial surgical treatment planning
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the sensitivity of the in vitro response of the organoid model to chemotherapeutic agents | 1 year
  Organoid treatment by means of ascending doses of chemotherapy and under HIPEC conditions, i.e. with elevated temperature
Next generation sequencing of organoid cultures | 1 year
  Sequencing of DNA and RNA (Ribonucleic acid)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Stange, Prof. Dr., Principal Investigator — University Hospital Carl Gustav Carus Dresden
Locations (2):
- Germany (2):
  - Department of Visceral, Thoracic and Vascular Surgery, University Hospital Carl Gustv Carus Dresden, Dresden
  - University Hospital Heidelberg, Heidelberg

IPD SHARING:
Plan to Share IPD: No